CLINICAL TRIAL: NCT03325335
Title: Randomized Controlled Trial Assessing the Effectiveness of Midazolam Premedication as an Anxiolytic, Analgesic, Sedative, and Hemodynamic Stabilizer
Brief Title: Assessing the Effectiveness of Midazolam Premedication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeon-Jeong Lee, Associate professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1607-003-057
Record Dates: First submitted 2017-10-22; First posted 2017-10-30 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Midazolam Premedication; Anxiety Preoperative; Premedication
Keywords: midazolam premedication
MeSH Terms: interventions — Transcobalamins; Remifentanil; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam premedication group (Group P) (Active Comparator): Patients of group P were premedicated with intramuscular midazolam 0.05 mg/kg 30 minutes before surgery.
  Interventions: Drug: Midazolam premedication; Drug: Remifentanil infusion; Drug: Propofol infusion
- Control group (Group N) (Other): Patients of group N were not premedicated with midazolam (Do not use placebo). [Treatment of Glycopyrrolate (0.2 mg, IM) 30 minutes prior to surgery is not intervention because it is a routine practice of this center. (-> removed from interventions)]
  Interventions: Drug: Remifentanil infusion; Drug: Propofol infusion

INTERVENTIONS:
Drug: Midazolam premedication — Patients in Group P received midazolam (0.05 mg/kg, intramuscular injection) 30 minutes before induction of general anesthesia.
  Other Names: Intramuscular midazolam
  Arms: Midazolam premedication group (Group P)
Drug: Remifentanil infusion — Target controlled infusion of remifentanil (4ng/ml) was used for induction of anesthesia based on the pharmacological models of Minto. After intubation, remifentanil (2 ng/ml) was infused until incision time. (Both groups)
  Other Names: Target-controlled infusion (TCI) of remifentanil
Drug: Propofol infusion — Target controlled infusion of propofol (4.0 μg/ml) was used for induction of anesthesia based on the pharmacological models of Marsh. After intubation, propofol (3.0μg/ml) was infused until incision time. (Both groups)
  Other Names: Target-controlled infusion (TCI) of propofol

SUMMARY:
Pre-anesthetic dosing of midazolam is commonly used in many hospitals for the induction of anesthesia, but the effect is still controversial. The purpose of this study was to evaluate the effectiveness of midazolam premedication in four aspects: anxiety reduction, pain relief, sedation and hemodynamic stability.

DETAILED DESCRIPTION:
Background

* Midazolam premedication is a routine practice in many hospitals, but its efficacy remains controversial. We evaluated the effectiveness of midazolam premedication with respect to anxiety and sedation levels, hemodynamic parameters, and analgesic profiles.

Methods

* Subjects

  * This randomized, prospective, open-label study was approved by IRB. After written informed consent, a total of 128 female patients aged between 20 and 65 years, ASA physical status Ⅰ or Ⅱ, scheduled for elective thyroidectomy were enrolled. Exclusion criteria were: central nervous system disorders, major cardiovascular disease, chronic pain disorders, peripheral neuropathy, diabetes mellitus neuropathy, nephropathy, hepatopathy, taking any medication affecting the central nervous system or heart rate, alcohol or drug abuse, pregnancy, and contraindication to midazolam premedication. Enrolled all subjects were randomly allocated to either midazolam premedication group (Group P, n=64) or control group (Group N, n=64). Patients of group P were premedicated with intramuscular glycopyrrolate 0.2mg and midazolam 0.05 mg/kg 30 minutes before surgery, while patients assigned to Group N were only received glycopyrrolate.
* Anesthetic management

  * In the operating room, we did standard monitoring(ECG, pulse oximetry, noninvasive blood pressure, esophageal stethoscope temperature), train of four (TOF) and entropy and surgical pleth index(SPI). Target controlled infusion of propofol (4.0 μg/ml) and remifentanil (4 ng/ml) were used for induction of anesthesia based on the pharmacological models of Marsh and Minto, respectively. Intravenous rocuronium 1.0 mg/kg was administered for muscle relaxation. After intubation, propofol (3.0μg/ml) and remifentanil (2 ng/ml) were infused until incision time. 30 mg of ketorolac was administered 30 minutes before the end of the operation to control postoperative pain.
* Assessment of response to midazolam

  * To evaluate the degree of anxiety, the Beck anxiety inventory was conducted at the preoperative day before surgery and immediately after arrival at the operating room. For analgesic profile assessment, SPI monitoring was performed in the operating room and NRS (numeric rating scale) measured in the recovery room and the general ward until the transition to oral analgesics. Also, additional medications for pain control were reviewed. Noninvasive blood pressure, heart rate, and entropy value were recorded at each measuring points in order to evaluate the hemodynamic stability and sedation level during anesthesia induction. Measuring points were initial time, prior to intubation, intubation, prior to incision and incision time. The time taken to induce anesthesia was also recorded.
* Sample size and statistical analysis

  * In this study, sample size was determined based on Cohen's study. According to this analysis, when comparing the mean of two groups with α (significance criterion) = 0.05, β (probability of occurring type II error) = 0.2 and medium effect size (Cohen's d = 0.5), 64 subjects were needed per group.
  * After a normality test, continuous variables were analyzed with the use of an independent t-test, paired t-test, and repeated-measures ANOVA. Differences between categorical variables were calculated with the use of the chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification I or II
* Scheduled for elective thyroidectomy under general anesthesia

Exclusion Criteria:

* Central nervous system disorders
* Major cardiovascular disease
* Chronic pain disorders
* Peripheral neuropathy
* Diabetes mellitus neuropathy
* Nephropathy
* Hepatopathy
* Taking any medication affecting the central nervous system or heart rate
* Alcohol or drug abuse
* Pregnancy
* Contraindication to midazolam premedication

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Change in degree of anxiety | the anesthesiologist's visit on the day before surgery and pre-induction time after randomization
  Patients completed the Beck anxiety inventory (BAI) on two separate occasions, the anesthesiologist's visit on the day before surgery and pre-induction time after randomization. The BAI was a self-report questionnaire consisting of 21 questions.
Change in sedation level | At the time of pre-induction (initial), prior to intubation, intubation, prior to incision, and surgical incision
  Measuring the entropy value (CARESCAPE Monitor B850, GE Healthcare, Milwaukee, WI, USA).
Change in noninvasive blood pressure (hemodynamic parameters 1) | At the time of pre-induction (initial), prior to intubation, intubation, prior to incision, and surgical incision
  Measuring noninvasive blood pressure (CARESCAPE Monitor B850, GE Healthcare, Milwaukee, WI, USA)
Change in SPI value (Analgesic profile 1) | At the time of pre-induction (initial), prior to intubation, intubation, prior to incision, and surgical incision
  Measuring SPI (CARESCAPE Monitor B850, GE Healthcare, Milwaukee, WI, USA), which was calculated from the pulse oximetry wave
Numeric rating scale (Analgesic profile 2) | Postoperative period (until transition to oral analgesics, up to 12 hours)
  Reviewing numeric rating scale (NRS) : 0 (No pain) ~ 10 (Worst possible pain)
Analgesic requirement (Analgesic profile 3) | Postoperative period (until transition to oral analgesics, up to 12 hours)
  Reviewing additional medications for pain control
Change in heart rate (hemodynamic parameters 2) | At the time of pre-induction (initial), prior to intubation, intubation, prior to incision, and surgical incision
  Measuring heart rate (CARESCAPE Monitor B850, GE Healthcare, Milwaukee, WI, USA)

SECONDARY OUTCOMES:
Procedure time of intubation | From the beginning of anesthesia to the completion of intubation
  Total time taken for intubation was recorded
Correlation analysis between the SPI values and other parameters (heart rate, blood pressure, and entropy values) | At the time of pre-induction (initial), prior to intubation, intubation, prior to incision, and surgical incision
  Measuring SPI, noninvasive blood pressure, heart rate, and entropy values (CARESCAPE Monitor B850, GE Healthcare, Milwaukee, WI, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Jeong Lee, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan national university hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No